CLINICAL TRIAL: NCT00002365
Title: A Randomized, Parallel, Open-Label Phase I Study of LXR015-1 in HIV-Infected Patients
Brief Title: A Study of LXR015-1 in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LXR Biotechnology (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 258A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-07

CONDITIONS: HIV Infections
Keywords: Dose-Response Relationship, Drug; Administration, Oral; Acquired Immunodeficiency Syndrome; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Drug: LXR015-1

SUMMARY:
To determine and compare the safety and tolerability of 3 doses of LXR015-1 in HIV-infected patients.

DETAILED DESCRIPTION:
Patients will be randomized to 1 of 3 doses of oral LXR015-1 for 28 days and patients will be monitored for adverse events for the duration of the study. Patients will continue to be monitored for least 4 weeks after completion of the dosing.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection.
* CD4 cell count less than 200 cells/mm3.

Prior Medication:

Allowed:

Acute therapy for opportunistic infections or serious AIDS defining infections must be completed at least 28 days before study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Patients that are unable to take adequate oral intake (i.e. unable to eat 1 or more meals a day because of chronic nausea, emesis, or abdominal/oral/esophageal discomfort).
* Patients who have severe diarrhea as defined as >= 7 stools per day, or acute diarrhea due to a treatable cause.

NOTE:

* If the patient has Cryptosporidia, Mycobacterium avium, or Cytomegalovirus that is unresponsive to treatment and has less than 7 stools per day, the patient may participate in this study.
* Patients who have any severe or life-threatening laboratory or clinical abnormality, or are not expected to live for 8 weeks.
* Patients who have an active opportunistic infection, including tuberculosis, cryptococcosis, or other serious AIDS defining infections requiring immediate treatment. Acute therapy must be completed at least 28 days before study entry.
* Patients with unexplained elevated temperature >= 38.5 degrees C that persists for 7 days or more within 14 days before study entry.
* Patients with malignancy other than squamous or basal carcinomas of the skin. Patients with visceral Kaposi's sarcoma or lymphoma requiring systemic chemotherapy or radiation treatment will be excluded. Patients with Kaposi's of the skin or mucous membranes may enroll in this study.
* Patients, who in the judgment of the investigator are unable to comply with the protocol.

Concurrent Treatment:

Excluded:

Radiation therapy.

Patients with the following prior condition are excluded:

A known history of hypersensitivity reaction to soy protein or soy lecithin. NOTE:

* This hypersensitivity is identified through medical history, not skin testing.

Excluded:

* Systemic chemotherapy.
* Acute therapy for opportunistic infections or other serious AIDS defining infections.
* Intravenous rehydration as treatment for diarrhea.

Required:

Patient must be taking a stable regimen (about 8 weeks) of anti-viral, anti-opportunistic infection and/or anti-diarrheal (if patient has diarrhea) medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Overall Officials: Bathurst I, Study Chair
Locations (1):
- East Bay AIDS Ctr, Berkeley, California, United States